CLINICAL TRIAL: NCT02295345
Title: Open Pilot of Cognitive Behavioural Therapy for Insomnia in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Lianne Tomfohr-Madsen, Assistant Professor of Psychology, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB14-0356
Record Dates: First submitted 2014-10-23; First posted 2014-11-20 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

ARMS (1):
- CBT for Insomnia (Experimental): Participants attend 5 weekly sessions of Cognitive Behavioural Therapy for Insomnia for pregnant women, administered by licensed clinical psychologist.
  Interventions: Other: Cognitive Behavioural Therapy for Insomnia

INTERVENTIONS:
Other: Cognitive Behavioural Therapy for Insomnia

SUMMARY:
Despite the literature showing cognitive behavioural therapy for insomnia (CBT-I) to be effective in a variety of populations including postpartum women, as well as the demonstrated harmful consequences of sleep disturbances in late pregnancy, no trials have investigated its efficacy during pregnancy. This project will investigate the efficacy and acceptability of cognitive behavioral therapy for insomnia (CBT-I) in pregnancy.

DETAILED DESCRIPTION:
Study details are included in the publication listed here: https://www.ncbi.nlm.nih.gov/pubmed/27124405

ELIGIBILITY:
Inclusion Criteria:

* English speaking women
* Over the age of 18
* Between twelve and twenty-eight weeks of gestation
* Identify as experiencing sleep disturbances will be recruited.

Exclusion Criteria:

* Women who identify as experiencing symptoms of sleep disorders other than insomnia (i.e. restless legs syndrome, obstructive sleep apnea)
* Women who are experiencing a current major depressive episode, or have been diagnosed with bipolar disorder or other disorders that have a psychotic, dissociative, hallucinatory, or delusional component
* Currently taking prescribed medications for sleep problems
* Inability to attend at least 4 out of the 5 weekly therapy sessions, participate in the assessments
* Smoking, drinking alcohol or drug use during pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Actigraphy indices from baseline to post-treatment | Baseline (Week 1), Post-treatment (Week 7)
  Actigraphy is recommended as a reliable and useful method of objective sleep assessment, providing information about indices of sleep efficiency, sleep latency, total sleep time, and number and frequency of awakenings
Change in Sleep Diary variables from baseline to post-treatment | Baseline (Week 1), Treatment (Weeks 2-6), Post-treatment (Week 7)
  Participants complete a daily, standardized sleep diary on a weekly basis both during the treatment period, and at baseline and final assessment times to corroborate actigraphy data. Dependent variables derived from this data include total sleep time, time in bed, sleep efficiency, and sleep quality
Change in Insomnia Severity Index (ISI) scores from baseline to post-treatment | Baseline (Week 1), Post-treatment (Week 7)
  The ISI can be used to assess the severity of sleep onset, sleep maintenance and early wakening problems, sleep dissatisfaction, and one's perceived distress caused by sleep problems. Scores on the ISI range from 0 to 28, with scores ≥ 15 indicating clinical insomnia.
Change in Pittsburgh Sleep Quality Index (PSQI) scores from baseline to post-treatment | Baseline (Week 1), Post-treatment (Week 7)
  The PSQI instrument is used in assessing one's sleep quality in the preceding month. It is comprised of 19 self-rated items and 5 questions rated by the roommate or bed partner. The PSQI possesses seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. PSQI scores range from 0 to 21, with scores greater than 5 indicating poor sleep quality.

SECONDARY OUTCOMES:
Change in Edinburgh Postpartum Depression Scale (EPDS) scores from baseline to post-treatment | Baseline (Week 1), Post-treatment (Week 7)
  The EPDS serves as a valuable and efficient way of identifying women at risk for prenatal depression, and can be used for screening both anxiety and depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of Calgary
Locations (1):
- University Of Calgary, Calgary, Alberta, Canada